CLINICAL TRIAL: NCT00995553
Title: Remediation of Working Memory in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Veterans Medical Research Foundation (Other); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6981-R; 1I01RX000180-01 (NIH)
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Remediation (Experimental): A 48-session working memory focused cognitive remediation program is conducted. Training tasks have been selected from 3 software programs, PSS CogRehab, BrainTrain, and custom made N-back tasks.
  Interventions: Behavioral: Cognitive Remediation
- Computer Skills (Placebo Comparator): This is a 48-session, time matched comparison group in which participants practice keyboarding skills and the fundamentals of Microsoft Office Word, Powerpoint, and Excel programs.
  Interventions: Behavioral: Computer Skills

INTERVENTIONS:
Behavioral: Cognitive Remediation — This is an adaptive, computer-based cognitive training intervention. Participants will complete 3 1-hour cognitive training sessions focused on attention and working memory processes weekly for 4 months.
  Arms: Cognitive Remediation
Behavioral: Computer Skills — This is a computer-based course in which participants will be taught how to use Microsoft Office applications and typing skills. Participants will attend a 1-hour course three times a week four 4-months.
  Arms: Computer Skills

SUMMARY:
The primary aim of the study is to test the efficacy of a novel cognitive remediation intervention that targets working memory-related functions. To accomplish this goal, 80 volunteer patients with schizophrenia will be enrolled and randomized to either a cognitive remediation condition that targets working memory or a computer skills training intervention that teaches computer applications. In both conditions participants will receive computer training three times a week for 4 months. The investigators hypothesize that patients who receive the cognitive remediation intervention will demonstrate significantly greater change on neuropsychological measures of working memory and executive abilities than patients who receive the computer skills course. In addition, the investigators hypothesize that the intervention-induced cognitive change will be associated with concurrent improvements in functional capacity and psychosocial functioning in the community. A second study goal is to examine the stability of the intervention-induced changes in cognition. Cognition and psychosocial functioning will be reassessed 4 and 8 months after treatment termination to examine the stability of treatment effects and to assess whether a less intense maintenance training (once a week sessions) provides any additional benefit to participants. Lastly, this study will examine in an exploratory manner whether there are individual differences in treatment response. The Val158Met polymorphism of the COMT gene has been found to be associated with working memory and prefrontal dysfunction in schizophrenia. The study will test whether the COMT polymorphism is predictive of response to cognitive remediation.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with a DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* No hospitalizations in the previous 4 weeks
* No antipsychotic medication changes in the previous 4 weeks
* Age 18-60
* Does not meet DSM-IV criteria for substance dependence in the previous 6 months or substance abuse in the previous month

Exclusion Criteria:

* History of clinically significant head injury or neurological disease
* Poor comprehension of the English language
* History of diagnosis of mental retardation or pervasive developmental disorder
* Unable to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2010-01; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tasha Marie Nienow, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Ramsay IS, Nienow TM, Marggraf MP, MacDonald AW. Neuroplastic changes in patients with schizophrenia undergoing cognitive remediation: triple-blind trial. Br J Psychiatry. 2017 Mar;210(3):216-222. doi: 10.1192/bjp.bp.115.171496. Epub 2017 Feb 2. PMID 28153927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 86 individuals were enrolled in the study. However, prior to condition assignment, 3 participants indicated that they needed to withdraw due to transportation problems, 1 participant withdrew due to a medical condition, and 1 participant lost interest in the study. Therefore, 81 participants were randomized to a study condition.
Period: Overall Study
Arm/Group | Cognitive Remediation | Computer Skills
Started | 40 | 41
Completed | 38 | 35
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Remediation | Computer Skills | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.83 (9.08) | 46.73 (10.24) | 46.28 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 33 | 28 | 61
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Assessment - MATRICS Consensus Cognitive Battery
Description: The Working Memory and Attention indexes of the MATRICS Consensus Cognitive Battery was used to assess near generalization of training with untrained tasks that were conceptually similar to training tasks. Each scale provide an age and gender corrected T-score. Thus, scores can range from 0-100, with a higher score indicating better performance.
Time Frame: Post-intervention, within 2 weeks of completion of the 4 month intervention
Population: All participants who engaged in the intervention, defined as completing at least 3 sessions, were included in an Intent to Treat analysis. 80 of the 81 participants who started one of the study conditions met this definition of engagement. One participant who attended only 1 session of computer skills was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cognitive Remediation | Computer Skills
Number analyzed (Participants) | 40 | 40
T-score
  MATRICS Working Memory Index | 40.08 (11.95) | 43.28 (11.80)
  MATRICS Attention Index | 39.80 (10.82) | 41.28 (10.11)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Computer Skills; MATRICS Working Memory Index; Test type: Superiority or Other; p = .06, ANOVA
Statistical Analysis 2: Comparison: Cognitive Remediation vs Computer Skills; MATRICS Attention Index; Test type: Superiority or Other; p = .09, ANOVA

2. Secondary Outcome: Functional Capacity - University of California, San Diego Performance-Based Skills Assessment
Description: The UPSA is a measure of the ability to apply cognitive skills to functional tasks. The total score from this scale was used. Scores may range from 0 - 100, with higher scores being better.
Time Frame: Post-intervention, within 2 weeks of completion of the 4 month intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation | Computer Skills
Number analyzed (Participants) | 40 | 40
units on a scale | 79.03 (10.60) | 78.78 (10.29)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Computer Skills; Test type: Superiority or Other; p = .73, ANOVA

ADVERSE EVENTS:
Arm/Group | Cognitive Remediation | Computer Skills
Serious Adverse Events (participants affected / at risk) | 7/40 | 7/41
Other Adverse Events (participants affected / at risk) | 3/40 | 3/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Remediation (N=40) | Computer Skills (N=41)
Hospitalization (Psychiatric disorders) | 7 (15) | 7 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Remediation (N=40) | Computer Skills (N=41)
Temporary symptom increase not requiring hospitalization (Psychiatric disorders) | 3 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No